CLINICAL TRIAL: NCT01455805
Title: Efficacy and Quality of Life Following Treatment of Lumbar Spinal Stenosis, Spondylolisthesis or Degenerative Disc Disease With the Minuteman Interspinous Interlaminar Fusion Implant Versus Surgical Decompression
Brief Title: Minuteman Spinal Fusion Implant Versus Surgical Decompression for Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Simplicity LLC (Industry)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SS2011UK
Record Dates: First submitted 2011-10-13; First posted 2011-10-20 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Lumbar Spinal Stenosis; Spondylolisthesis; Degenerative Disc Disease
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis; Intervertebral Disc Degeneration | interventions — Decompression, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minuteman Fusion Implant (Active Comparator): Minuteman™ interspinous interlaminar fusion Implant (interspinous interlaminar fusion device) which gained CE Mark approval in May 2011
  Interventions: Device: Minuteman Fusion Implant
- Surgical decompression (Other): Surgical decompression refers to the following operations Laminectomy, Foraminotomy, Discectomy or any other surgical procedure that the clinician feels is relevant for the decompression of lumbar spinal stenosis.
  Interventions: Procedure: surgical decompression

INTERVENTIONS:
Device: Minuteman Fusion Implant — The Minuteman™ interspinous interlaminar fusion device consists of a central threaded portion that has a two-part wing plate hinged near its proximal end, with spikes on the extended distal end of the wing plate, and a multi-spiked end cap plate that is located at the distal end of the device and is retained and tightened in place with a locking hex nut. Compression between the spiked wing plate and the spiked end cap plate serves to fix the spinous processes in place and to facilitate fusion, together with bone graft fusion material placed within the device. The threaded external body has been designed to provide ease of distraction and insertion via a minimally invasive surgical procedure.
  Other Names: The Minuteman™ interspinous interlaminar fusion device
  Arms: Minuteman Fusion Implant
Procedure: surgical decompression — Surgical decompression refers to the following operations Laminectomy, Foraminotomy, Discectomy or any other surgical procedure that the clinician feels is relevant for the decompression of lumbar spinal stenosis
  Arms: Surgical decompression

SUMMARY:
Lumbar spinal stenosis (LSS), is a common disorder of narrowing of the spinal canal in the lower part of the back. This causes discomfort in the legs when standing or walking because of pressure on the spinal nerves.There are several treatment options for LSS including physiotherapy, lumbar surgical decompression procedures such as laminectomy, Foraminotomy, Discectomy and more recently devices for interspinous distraction such as the XSTOP® and from May 2011 Minuteman™.

Surgical decompression for LSS involves the removal of excess bone, ligament, and soft-tissue allowing more room for the nerves. The operation is usually preformed under general anaesthetic and with an average stay in hospital for 2-3 nights. Whereas the Minuteman™ implant is preformed as a day case under local or general anaesthetic and involves implanting the device into the space between two back bones to relieve pressure on the nerves and, therefore, pain in the legs.

This is a multi centred (four sites) randomised controlled trial with a total sample of 50 participants after obtaining their informed consent. Participants will attend the pain clinic at the Hospitals for a baseline visit where they will be randomised with a ratio of 1:1 to receive either the Minuteman™ Interspinous interlaminar fusion Implant or standard surgical decompression for the treatment of lumbar spinal stenosis (LSS). Following randomisation arrangements will be made for the participant to receive the randomised treatment. If allocated to Minuteman™ Implant, the treatment will be conducted by the Pain Specialist identified at the site. If allocated to surgical decompression, the treatment will be conducted by the neuro/spinal-surgeon identified at the site. Participates will be followed up regularly for 60 months post implant to assess clinical efficacy, safety, participants function and quality of life of each treatment.

DETAILED DESCRIPTION:
This is a prospective randomised study monitoring patients for up to 5 years post treatment. Only patients who have an appropriately diagnosed Lumbar Spinal Stenosis with intermittent claudication with/without low back pain, with no adequate symptomatic relief after at least 6 months of conservative treatment will be asked to give consent to be involved. Potential participants will be approached for enrollment 17days before the planned baseline visit. Patients will be given oral and written information about the trial as well as the patient information leaflet for the study. If informed consent is given their participation in this study will be for a maximum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Is male or a non pregnant female aged 18years or older
* BMI ≤ 35kg/m2
* Has chronic leg pain with or without back pain of greater than 6 months duration,which is partially or completely relieved by either sitting or adopting a flexed posture and who are suitable in the clinicians opinion for posterior lumbar surgery
* Pre-operative ODI score ≥ 20%
* Pre-operative ZCQ Physical Function Domain ≥2
* Pre-operative VAS Leg pain score ≥ 4
* Has completed at least 6 months of conservative treatment without obtaining adequate symptomatic relief or has worsening neurological symptoms.
* Has degenerative changes at 1 or 2 levels confirmed by MRI or CT Myelogram within the last 12 months) with one or more of the following:
* Lumbar spinal stenosis with intermittent neurogenic claudication
* Degeneration of the disc (as evidenced by imaging on MRI)
* Annular thickening
* Degenerative Spondylolisthesis ≤ Meyerding Grade 1
* Thickening of ligamentum flavum

Exclusion Criteria:

* Fixed motor deficit
* Has undergone previous lumbar spinal surgery
* Is unwilling or unable to give consent or adhere to the follow up schedule
* Has active infection or metastatic disease
* Has spondylolisthesis > grade 1
* Has neurogenic bladder or bowel disease
* Has a history of Osteopenia and or Osteoporosis. Evaluation of possible Osteopenia and or Osteoporosis will be conducted via a bone density scan prior to randomisation if ANY of the Bone Mass Evaluation criteria is met
* Patients who are not deemed fit for anaesthesia/major surgery due to underlying medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-06; Primary Completion 2024-03 (Actual); Study Completion 2024-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline of clinical efficacy up to 60 months post procedure | 8 weeks and up to 60 months post procedure.
  These include:
  * Visual Analogue Scale (VAS) pain scores Leg Pain
  * Visual Analogue Scale (VAS) pain scores Back Pain
  * Oswestry Disability Index (ODI)
  * Zurich Claudication Questionnaire (ZCQ)
  * Assessment of Physical Function via distance walked in 5 minutes and number of repetitions of sitting to standing in 1 minute.
  The main outcome will be a comparison between treatment groups based on the change from baseline at each follow-up visit for each of the measures listed above.

SECONDARY OUTCOMES:
measures of quality of life | 8 weeks and up to 60 months post procedure.
  These include:
  * Change in functional status questionnaire from baseline
  * Participants global impression of change from baseline (PGIC)
  * Clinician's global Impression of change from baseline (CGIC)
  * Employment status
Adverse events related to device and procedure | safety to be assessed at 8 weeks and up to 60 months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ganesan Baranidharan, Dr, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (4):
- United Kingdom (4):
  - Taunton & Somerset NHS Foundation Trust of Musgrove Park Hospital, Taunton, Somerset
  - The Ipswich Hospital NHS Trust, Ipswich, Suffolk
  - Pain and Interventional Neuromodulation Research Group, Pain Management Dept, Seacroft Hospital, Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire
  - The Dudley Group NHS Foundation Trust, Russell Hall Hospital, Birmingham